CLINICAL TRIAL: NCT04471090
Title: Effects of Positional Therapy on Pulmonary Physiology in Patients Undergoing Mechanical Ventilation.
Status: Completed | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Fernando Suarez Sipmann, MD PhD Intesive Care Medicine, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Other Study IDs: PT-IMV
Record Dates: First submitted 2020-07-01; First posted 2020-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this project is to evaluate the effects of positional changes in mechanically ventilated patients.

DETAILED DESCRIPTION:
In critically ill patients undergoing invasive mechanical ventilation (IMV), several negative effects converge, promoting the development of collapse in the dorsal areas of the lung. These among others include deep sedation, relaxation, prolonged immobility and the supine position. This results of an added impairment in lung function both in the mechanical and gas exchange. In addition lung collapse contributes to a significant increase in the heterogeneity the distribution of alveolar ventilation and perfusion that may increase the risk of ventilator-induced lung injury (VILI).

Postural therapy is widely recommended as prevention/treatment of pressure ulcers, whose presence, according to the Spanish Society of Intensive Care Medicine (SEMICYUC), is a quality criterion for intensive care units (ICUs), with a prevalence of 18% in these units compared to 7.8% in adult hospitalization. However, how postural changes may affect lung function is an aspect that has been scarcely studied. Given the strong influence of gravity on lung function, positional changes can produce significant alterations in the distribution of trans-pulmonary pressures (a decrease along the vertical gravitational axis of approximately 0.25 cmH2O per cm). Depending on the severity, distribution and location of the respiratory pathology, positional changes may have a significant effect either benefiting or impairing the patient's condition.

The investigators will dynamically assess the effects of routine lateral positioning up to 30-40º by means of electrical impedance tomography (EIT), a non-invasive, radiation-free functional bedside imaging technique that allows to monitor the regional distribution of ventilation and perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IMV under sedation, in a controlled ventilatory modality in passive conditions (i.e. without any spontaneous inspiratory efforts by the patient).
* Signature of the informed consent by family member or legal representative.

Exclusion Criteria:

* Presence of any clinical contraindication for postural therapy, including patient haemodynamic instability, traumatism, pathology or any other cause.
* Contraindication for the placement of the EIT electrode belt due to unstable spinal cord injury or other skin injuries or wounds in the thoracic region (surgical, traumatic, etc.)
* Assisted ventilatory modes in a non-passive breathing patient.
* Hypernatremia
* Patients with pacemakers or implantable automatic defibrillators (IAD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted in the ICU of La Princesa University Hospital, Madrid, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Regional ventilation and perfusion distribution ratio | 60 minutes
  Percentage of relative ventilation in each Region Of Interest (ROI) in each of the studied positions
Global mechanical compliance and regional impedance compliance | 60 minutes
  Global mechanical compliance and regional impedance compliance (CZ) for each ROI in each of the studied positions.

SECONDARY OUTCOMES:
Assessment of lung mechanics. | 60 minutes
  Changes in the lung mechanics during postural changes in their usual positions: supine position (SD), right lateral position (RLP) at 30º and left lateral position (LLP) at 30º. Global compliance and regional compliance (impedance arbitrary units/cmH2O)
Assessment of ventilation/perfusion lung distribution. | 60 minutes
  Changes in the regional distribution of lung ventilation and perfusion during postural changes in their usual positions: supine position (SD), right lateral position (RLP) at 30º and left lateral position (LLP) at 30º. Percentage of relative ventilation and perfusion distribution in each region of interest (ROI). Relative distribution (%) and derived indexes.
Assesment of changes in ventilation/perfusion in prone position. | 60 minutes
  Changes in ventilation and perfusion in prone position if during the study this circumstance arises due to medical indication. Percentage of relative ventilation and perfusion distribution in each region of interest (ROI). Relative distribution (%) and derived indexes.
Assessment of the effects of postural therapy in cases of predominantly unilateral lung pathology | 60 minutes
  Effects of postural therapy in cases of predominantly unilateral lung pathology. Percentage of relative ventilation and perfusion distribution in each region of interest (ROI). Relative distribution (%) and derived indexes.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Suarez Sipmann, MD PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de La princesa, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No